CLINICAL TRIAL: NCT06525129
Title: Comparison of Multi-session Anodal Cerebellar Transcranial Direct Current Stimulation vs Anodal Cerebral Transcranial Direct Current Stimulation on Balance, Its Components and Postural Stability in Stroke Patients
Brief Title: Multi-session Anodal Cerebellar Transcranial Direct Current Stimulation (tDCS) vs Anodal Cerebral tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Qurat ul Ain3
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cerebellar stimulation group (CbSG) (Experimental)
  Interventions: Other: Cerebellar stimulation group (CbSG)
- Cerebral (M1) Stimulation group (MSG) (Experimental)
  Interventions: Other: Cerebral (M1) Stimulation group (MSG)
- Sham Stimulation group (SSG) (Other)
  Interventions: Other: Sham Stimulation group (SSG)

INTERVENTIONS:
Other: Cerebellar stimulation group (CbSG) — Anodal transcranial direct current stimulation was given using a portable battery-driven brain stimulator (The Brain Stimulator v3.0 Deluxe tDCS Kit, using Professional 3x3 inches Amrex Sponge Electrodes). Skin was prepared before application of electrodes by cleaning the skin surface using alcohol swabs. In cerebellar stimulation group (CbSG) a stimulation intensity of 2mA for duration of 20 minutes. In order to avoid sudden initiation and termination of the stimulation the first and last 10 seconds of anodal tDCS application, current will gradually fade in/fade out to avoid any sudden starting or stopping of the stimulation. For the CbSG active anodal electrode was placed over the cerebellum with about 1-2 cm below inion occipital protuberance, whereas the returning cathodal electrode was placed on right buccinator muscle.
  Arms: Cerebellar stimulation group (CbSG)
Other: Cerebral (M1) Stimulation group (MSG) — In the M1 Stimulation Group (MSG) a similar intensity of current with 2mA was applied for a period of 20 minutes. Skin was cleaned with alcohol swab ahead of placing the electrodes. The anode was positioned over the lesioned M1 motor cortex area (C3, International 10-20 system) while the cathode was placed over the contra-lateral supraorbital area. Due to the large size of electrodes, the active electrode covered the area of M1 for the hand, arm, trunk, and the LL. Ten sessions of anodal tDCS were applied over a duration of 2 weeks. The stimulation was applied during active participation of patients in Biodex balance training.
  Arms: Cerebral (M1) Stimulation group (MSG)
Other: Sham Stimulation group (SSG) — In Sham Stimulation group (SSG) Ten sessions of anodal tDCS were applied over a duration of 2 weeks having same intensity i.e., 2 mA stimulation was used for a period of 30 seconds and then gradually ramped-down and turned off for the rest of the treatment time of 20 minutes. The same procedure for skin preparation was used as in the other two groups. Electrode placement for SSG was same as in MSG for half of the patients i.e. 8 participants; anode will be placed over the left (dominant) lesioned M1 whereas the cathode will be positioned over the right (contralateral) supraorbital area. For the other 8 participants the stimulation montages were similar to cerebellar stimulation group. The active anodal electrode was placed over the cerebellum with about 1-2 cm below inion occipital protuberance, whereas the returning cathodal electrode was placed on right Buccinator Muscle.
  Arms: Sham Stimulation group (SSG)

SUMMARY:
To investigate which one of the two cerebellar and cerebral stimulation in comparison to sham stimulation is more effective in enhancing balance and postural stability in stroke patients

ELIGIBILITY:
Inclusion Criteria:

* The study focused on individuals who had their first stroke,
* Additionally, participants needed to have a score of 6 or higher on the Johns Hopkins Fall Risk Assessment Tool (JHFRAT).
* The inclusion criteria mandated that participants must have the ability to give written consent, walk without any help, and
* have a functional condition that allows them to actively participate in the Biodex balancing training program.

Exclusion Criteria:

* Individuals with concurrent neurological problems such as Alzheimer's, Parkinson's, or cerebellar abnormalities,
* as well as those with psychological ailments, were excluded during the initial assessment phase.
* In addition, individuals who scored below 20 on the Mini Mental Status Examination Test (MMSE),
* displayed motor disorders that affected their ability to walk or use their lower limbs,
* were currently taking sedative medications, had amnesia, depression, radiculopathy, lumbar spinal cord root involvement, auditory or visual impairments, vertigo, recent fractures, severe cardiac problems,
* or had undergone electrotherapy that affected their nervous system within the past two weeks were also not included in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Biodex balance system | 2 weeks
  The biodex balance system based specific dynamic postural tests were delineated for implementation on both static and dynamic levels. Postural stability tests were performed at three levels of stability: 12 (maximum stability = static), 7 (moderate stability) and 3 (slight stability).
Berg balance scale | 2 weeks
  The Berg balance scale (BBS) is used to assess the participant's ability to retain stability.
  The BBS is a widely used test for the assessment of the elderly population with impairment of balance and individuals with neurological disorders while sitting, standing, and transferring. This test included both static and dynamic type tasks. The BBS uses a five-point ordinal scale ranging from 0 (disability) to 4(complete independent performance) and consists of 14 components; the maximum score is 56 points. The scale has been shown to be reliable and valid in stroke patients. A cut-off score of 45 points is used for fall prediction. The BBS involves 14 tasks: a total score of 56. Equipment required for this test was a stopwatch or watch with a second hand and a ruler or other indicator of 2, 5, and 10 inches.
Timed up and go test | 2 weeks
  The Timed Up and Go (TUG) test was designed for the evaluation of balance and Measures mobility in people who are able to walk on their own (assistive device permitted) to find out the risk of fall. The subjects will be required to stand up from a chair, walk 3 m, turn around, return to the chair, and sit down. The time taken to complete this task will be measured. The test will be informed three times. The time required to complete this task will be measured from a stopwatch. The average values from 3 trials, with 1-min rest between each trial, were used for data analysis.
Bestest balance evaluation system | 2 weeks
  Changes from the base line, immediately after Intervention and then again after 1 hour.
  Balance Evaluation Systems Test (BESTest) is a 36-item assessment of balance impairments across 6 postural control contexts. Total score of 108 points total, calculated into a percentage score (0-100%). Also, total sub-scores exist for each above listed system. Item- level scores range from 0 (severe impairment) to 3 (no impairment)
TDCSs adverse effects questionnaire | 2 weeks
  Transcranial Direct-Current Stimulation (tDCS) adverse effects questionnaire:
  Do you experience any of the following symptoms or side- effects? Headache, Neck pain, Scalp pain, Tingling, Itching, burning sensation, Skin redness, Sleepiness, Trouble concentrating, Acute mood change, Others (specify) for each symptom patient can give value (1-4) (1, absent; 2, mild; 3, moderate; 4, severe). If present: Is this related to tDCS?
  (1, none; 2, remote; 3, possible; 4, probable; 5, definite)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Study Chair — Riphah International University; Qurat Ul Ain, PhD*, Principal Investigator — Xi'an Jiaotong University
Locations (1):
- Akbar Hospital, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No